CLINICAL TRIAL: NCT07103044
Title: Developing Early Achievements for Pre-K Children With Developmental Language Disorders: A Comprehensive Contextualized Embodied Approach
Brief Title: Early Achievements - Shaping Early Language and Literacy Skills
Acronym: EA-SHELLS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: Institute of Education Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00294058; R324A210031 (Other Grant/Funding Number: Institute of Educational Sciences)
Record Dates: First submitted 2025-07-10; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Developmental Language Disorder
Keywords: Literacy; Reading; Language; Education
MeSH Terms: conditions — Language Development Disorders; Literacy; Language

STUDY DESIGN:
Intervention Model Description: Upon confirmation of eligibility and completion of the baseline assessments, teachers will be randomly assigned to the Full Training group or the Quick Training group. Randomization will be done at the classroom level as teachers will implement the instructional approach with their whole class rather than specific students.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Full Training Group (Experimental): Teachers assigned to the Full Training group will participate in a collaborative coaching approach, Practice-Based Coaching (Snyder et al., 2015). Coaches will support teachers in targeting meaning-related (language-based) emergent literacy skills during whole and small group interactions with their students. The duration of the coaching period is approximately 14 weeks with about one coaching session per week. Teachers will be coached to implement Early Achievements-Shaping Early Language and Literacy Skills (EA-SHELLS) strategies during book reading and book-related activities. See more details about the instructional approach below in the intervention description.
  Interventions: Behavioral: Early Achievements - Shaping Early Language and Literacy Skills
- No Intervention: Quick Training Group (No Intervention): Teachers assigned to the Quick Training group will not receive any training or intervention while data are being collected from both groups. Teachers in this group will conduct their classroom instruction as originally planned while the teachers in the Full Training group receive the EA-SHELLS training. After the completion of data collection, teachers will be invited to participate in a collaborative coaching approach, Practice-Based Coaching (Snyder et al., 2015). Coaches will support teachers in targeting meaning-related emergent literacy skills during whole and small group interactions with their students for 2 coaching sessions. Teachers will be coached to implement EA-SHELLS strategies during book reading and book-related activities. Teacher data will be collected during the quick training period but will be analyzed separately from RCT data used to examine efficacy of EA-SHELLS.

INTERVENTIONS:
Behavioral: Early Achievements - Shaping Early Language and Literacy Skills — EA-SHELLS is a professional development program that includes a 6-hour workshop and about 14 in-person coaching sessions using Practice-Based Coaching. Teachers will implement the EA-SHELLS instructional approach in their classrooms during whole-group book sharing activities to target vocabulary, syntax, story grammar, and listening comprehension. Teachers will also lead story retelling activities using pictures cards and 3D props to further target all four skills. Teachers will be provided with commercially available children's books augmented with supplemental text to explicitly define vocabulary and cue teachers' elicitation of children's verbal engagement for targeted vocabulary, syntactically elaborated sentences, and story grammar elements. Instructional strategies include naturalistic developmental behavioral intervention and language facilitating (e.g., focused stimulation) strategies. Teachers will read each provided book about four times over one to two weeks.
  Arms: Experimental: Full Training Group

SUMMARY:
Language skills are important for long-term reading comprehension success. Yet there are limited instructional approaches available for prekindergarten (pre-K) teachers to use in their inclusive classrooms to boost literacy-related language skills in children with and without language delays or disorders.

In the first part of this study, the investigators will develop a teacher training program focused on building pre-K children's language-based literacy skills. Teachers will be trained and will use the strategies that they learn during literacy-related activities in their inclusive pre-K classrooms. Their students' language-related literacy skills will be measured before and after their training. Based on teacher feedback and child assessment information, the training program will be revised. In the final part of the study, a preliminary randomized control trial (RCT) will be done using the revised training approach. The results of the RCT will help the investigators know if the teacher training program helps to improve the effectiveness of teachers' instruction and their students' development of language-related literacy skills.

The primary goal of this research study is to determine whether study-trained pre-K teachers in inclusive early childhood education classrooms use more effective teaching strategies than teachers who do not receive the training. A secondary goal of this research study is to determine if this teacher training program strengthens language-related literacy skills for students with and without language disorders or delays. The research team hypothesizes that teachers who participate in the training program will use effective teaching strategies more often than teachers who do not receive the training. Additionally, the investigators predict that teachers who receive the training will feel more confident teaching early language-based literacy skills to their students (with and without language delays/disorders) than teachers who do not receive the training. Researchers also predict that students taught by teachers who receive the training will perform better on language tests when compared to their peers in classrooms where the teacher training program was not used.

DETAILED DESCRIPTION:
The primary goal of this research study is to determine whether Early Achievements - Shaping Early Language and Literacy Skills (EA-SHELLS) training improves teachers' implementation of the EA-SHELLS instructional approach in their inclusive prekindergarten (pre-K) classrooms. A secondary purpose of this research study is to determine the effects the EA-SHELLS instructional approach on pre-K children's (with and without language disorders/delays) language-related emergent literacy skills (vocabulary, syntax, narrative representation, and listening comprehension). The investigators hypothesize that teachers who participate in the EA-SHELLS professional development program will show greater use of evidence-based instructional strategies (the EA-SHELLS approach) and greater self-efficacy relating to language-related literacy instruction compared to teachers who do not receive the training. Additionally, the investigators predict that students taught by teachers receiving the training will perform better on testing measures when compared to their peers who do not receive supported classroom instruction.

An iterative development process was utilized for this study. Phase 1 (initial development and implementation) and Phase 2 (iterative development and implementation of the intervention) took place prior to this clinicaltrials.gov submission. A total of 17 teachers and 87 students completed the full research program in these phases. Preliminary results show significant positive outcomes on student and teacher measures.

In Phase 3 (randomized control trial), investigators will further test the above hypotheses by collecting data from teacher and student participants at pre-treatment, midpoint, and post-treatment time points in comparison to teachers and students who do not receive the training. The duration of the study will last approximately 14 weeks. Teachers may be randomly assigned to receive either the full training or no training until after post-treatment data are collected. Teachers in the EA-SHELLS trained group will attend the 6-hour virtual EA-SHELLS workshop and participate in approximately 14 in-person coaching sessions. During this EA-SHELLS training period, data will be collected on teacher and student participants in both arms of the trial.

ELIGIBILITY:
Inclusion Criteria for Teachers

* Having students in the identified age range
* Having at least one child in their classroom who receives language-focused related services, has an existing diagnosis of language delay or disorder, or meets study criteria for DLD on the research measures
* Planning to teach for the duration of the training period.

Inclusion Criteria for Students in the DLD group:

* use phrases containing a noun and a verb in most spontaneous utterances (per teacher report)
* are exposed to English >50% of their time at home (per parent report). receive language-focused related services, have a prior diagnosis of language delay or disorder, or meet study criteria for language delay on the CELF P-3 and/or CUBED NLM.
* CELF P-3: score more than 1 standard deviation below the mean on at least one subtest
* NLM criteria: receives two Listening Retell score raw score of <5 on Fall measures or <7 on Winter measures
* between approximately 45-65 months of age

Inclusionary criteria for students in the TD group:

* cannot have an identified DLD or developmental disability and does not meet above criteria for language delay/disorder
* between approximately 45-65 months of age.
* are exposed to English >50% of their time at home (per parent report)

Exclusion Criteria:

Exclusionary criteria for both the DLD group and TD group:

* having a visual or hearing impairment after correction (per parent report)
* having a motor impairment that renders them unable to reach and grasp objects or sit independently
* score more than1.5 standard deviation below the mean on the Mullen Scales of Early Learning Visual Reception subscale
* This criterion will be evaluated on a case-by-case basis at the PI's discretion as children's performance may be affected by any of a number of factors and a single response variation may result in a child missing the cut-off while clearly succeeding cognitively in the classroom.

Ages: 45 Months to 65 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2021-08-26 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of Story Comprehension (ASC) | Baseline and post 14-week training period
  This measure serves as an indicator of narrative comprehension at pre- and post-treatment time points. Students will be administered two parallel versions of this assessment at both testing points. The combined raw score will be used for comparison. This measure was used in iterative development phases and will be used in the RCT
Narrative Language Measure - Listening (NLM) | Baseline
  This measure serves as an indicator of narrative comprehension at pre- and post-treatment time points. Students will be administered two parallel versions of this assessment at both testing points. The combined raw score will be used for comparison. This measure was used in iterative development phases and will be used in the RC
Vocabulary Assessment | Baseline and post 14-week training period as well as every 2-4 weeks during the training period.
  This researcher created measure assesses vocabulary learning throughout the study. Students will participate in testing at pre- and post-treatment time points. Additionally, students will participate in monthly intra-intervention testing. Raw scores will be used for data analyses. This measure was used in iterative development phases. It was revised across phases. The most updated version will be used in the RCT.
The Narrative Assessment Protocol-Second Edition (NAP-2) | Baseline and post 16-week training period
  This measure was used in early iterative phases to measure syntax and narrative production, without transcription. Two stories were used (equated on length and difficulty) each at pre-, mid-point and post-treatment (constant across children and phases), with one story given at all three times to control for confounding effects of different stories administered per the authors' recommendation.
Expressive Vocabulary Test, Third Edition (EVT-3; Williams, 2019) | Baseline (served as a participant characterization measure).
  This student assessment was used in early iterative phases of this research. It was used as a direct assessment of generalized expressive vocabulary performance. This measure will not be used in the RCT.

SECONDARY OUTCOMES:
Clinical Evaluation of Language Fundamentals - Preschool, 3rd Edition (CELF-P3) | Baseline and post 14-week training period
  This measure serves as an indicator of overall language ability at pre- and post-treatment time points. Additionally, this test helps differentiate between TD and DLD students. Students will be administered the following subtests: Sentence Comprehension, Word Structure, Expressive Vocabulary, and Basic Concepts. This measure was used in iterative development phases and will be used in the RCT.
Teacher Book and Book-Related Activity Fidelity | Baseline and post 14-week training period as well as 1-3 times during the training period
  Video recordings are collected and coded (masked to group and timepoint) to evaluate teachers' implementation fidelity of book and book-related activities in their classrooms. Videos will be collected pre- and post-treatment as well as approximately 1-3 times during the training period (intra-intervention). These measures were used in iterative development phases and will be used in the RCT.
Teacher Satisfaction and Feasibility Survey | Post 14-week training period.
  This survey provides insights about EA-SHELLS features that inspire willingness to use and those that present implementation barriers and/or facilitators (related to feasibility). A subset of items addresses perceptions of the feasibility and satisfaction of EA-SHELLS, as will open-ended questions about how to improve each component of EA-SHELLS to engage and enrich learning for their students. Data collected from iterative development phases was used to inform revisions to maximize practicality of adopting the intervention. This measure will continue to be used in the RCT to measure satisfaction with, and perceptions of, the feasibility of EA-SHELLS.
The Barriers Checklist | Post 14-week training period.
  This survey was adapted from Bartholomew et al. (2007) and consists of 10 items pertaining to resources (e.g., insufficient time, resource, training) and procedural barriers (e.g., complexity, compatibility) that threaten usability and feasibility. This measure was used in iterative development phases to inform revisions to the intervention. We will continue to use this measure in the RCT to provide information regarding teacher perceived barriers to implementation of EA-SHELLS.
The Teacher Consumer Review Form | Post 14-week training period.
  This survey is a 5-point Likert-type scale to rate EA-SHELLS components (scope and sequence, instructional contexts, instructional strategies, materials, and PD) regarding: (1) relative advantage over currently available (or previously experienced) oral language interventions (including cost); (2) compatibility with available resources and organizational structures, work demands, and instructional practices already used; and (3) complexity of the content, activities, and structure of the intervention. For each dimension, teachers are asked to describe two ways to improve the program to increase its relative advantage and overall compatibility, and to reduce complexity. This measure was used in iterative development phases and will be used in the RCT.
The Self-Efficacy Scale | Post 14-week training period.
  This survey is completed by teachers at pre- and post-treatment to document their confidence in delivering the EA-SHELLS intervention. Results will have implications for the usability and feasibility of EA-SHELLS and perceived complexity. During the iterative development phase, this scale was given to all teacher participants. Responses influenced revisions to the intervention. For the RCT, this scale will only be given to teachers in the Full Training group.
Teacher Self-Rating of Coaching Impact | Post 14-week training period
  This researcher developed survey provides information about the social validity, feasibility, and practicality of the coaching process and content obtained. This measure was used in iterative development phases and will be used in the RCT.
Adapted Texas Christian University Workshop Evaluation Form | Baseline, after the initial workshop training.
  Researchers adapted the Texas Christian University Workshop Evaluation Form (Institute of Behavioral Research, 2002) to address a DLD and TD populations included in this study. This survey consists of 22 items each rated on a 5-point Likert-type scale. Data collected measure teachers' reactions to workshop content and intentions to implement EA-SHELLS components. This measure was used in iterative development phases and will be used in the RCT.
Demographic Forms | Baseline
  Demographic information is collected for both student and teacher participants. Data is collected via an online survey. Teachers provide additional information regarding education and teaching experience. Surveys focused on children include specific questions regarding development and any diagnosed developmental delays. These measures were used in iterative development phases and will be used in the RCT.
EA-SHELLS Home Survey | Baseline
  The EA-SHELLS Home Survey is a researcher created measure relating to participants' exposure to books and early literacy/communication enhancing strategies at home. The Home Survey consists of 15 multiple choice and Likert scale items. This measure was used in iterative development phases and will be used in the RCT.
Teacher Rating of Oral Language and Literacy (TROLL), adapted | Baseline
  Teacher participants complete an adapted version of the TROLL (Dickinson et al., 2003) for each consented student. This teacher completed survey provides information pertaining to students' language and literacy skills as observed by their teacher in their daily classroom routines. This measure was used in iterative development phases and will be used in the RCT.
Focus Group Feedback | Baseline and post 14-week training period
  Focus group meetings last approximately 1 hour and use a set of IRB approved interview questions. Teacher responses are transcribed and qualitatively analyzed. This measure was used in iterative development phases and will be used in the RCT. In iterative development phases, all teacher participants attended pre- and post-training focus group meetings. In the RCT, only teacher participants in the Full Training Group will attend pre- and post-treatment focus group meetings.
Unit Review Forms | Every 2-4 weeks throughout the training period
  Teachers complete the researcher-created forms at the end of each intervention unit. Teachers report the frequency with which they use instructional strategies as well as their perceived strengths and challenges when instructing their students. This measure was used in iterative development phases and will be used in the RCT.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Landa, PhD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger Institute
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: This page provides an overview of the EA-SHELLS study for interested teachers to learn more about participation. — https://www.kennedykrieger.org/training/programs/ea-shells